CLINICAL TRIAL: NCT01897818
Title: Communication by Brain - Computer Interface in Amyotrophic Lateral Sclerosis:Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-PP-16
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-05

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

ARMS (1):
- ALS patients (Experimental)
  Interventions: Device: communication system P300 Speller

INTERVENTIONS:
Device: communication system P300 Speller

SUMMARY:
ALS is a severe progressive neurodegenerative disease characterized by degeneration motor neurons leading to death in 3 to 5 years. Gradually in time, the patient deprived of all motor skills as well as the possibility of communication written and oral developing a state close Locked In Syndrome (LIS). The main objective is to establish the feasibility of brain-computer interface using the pathological condition, with dependent disabled subjects as a means of communication.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18
* have a diagnosis of ALS suspected, possible, probable with EMG
* be able to follow the study process and to comply with the schedule of visits upon entry into the study
* understand the purpose of the study
* expressing P300 wave in the conditions of the study

Exclusion Criteria:

* have a mental illness or clinical dementia defined clinically significant may hinder the patient's ability to follow the procedures of the study
* have a significant history of photosensitive epilepsy
* have a history of allergy to the gel used for the electrodes
* Major protected by law (guardianship, curators)
* have uncorrectable visual disorders
* not being able to maintain a sitting position and focus on a computer screen for more than 30 min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-07; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
the full achievement of "copy spelling" and "free spelling" tests session 1 | 14 days after inclusion
the full achievement of "copy spelling" and "free spelling" tests session 2 | 28 days after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de l'Archet I, Nice, France